CLINICAL TRIAL: NCT03471897
Title: Plasma Glycosaminoglycans as Diagnostic and Prognostic Biomarkers in Surgically Treated Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Chalmers University of Technology (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: GAG-RCC-03
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Renal Cell Carcinoma
Keywords: glycosaminoglycans; biomarkers; diagnostics; prognostic; liquid biopsy
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RCC: Patients with pathologically confirmed diagnosis of RCC
  Interventions: Diagnostic Test: Glycosaminoglycan plasma score
- Controls: Subjects self-reported as healthy
  Interventions: Diagnostic Test: Glycosaminoglycan plasma score

INTERVENTIONS:
Diagnostic Test: Glycosaminoglycan plasma score — A score was calculated using a formula that factors in measurements of plasma glycosaminoglycan. A score higher than a here-determined threshold is deemed diagnostic of RCC.

SUMMARY:
In this study, the investigators profiled plasma glycosaminoglycans (GAGs) in a retrospective consecutive series of patients with a radiographic finding of renal mass referred to primary surgery for renal cell carcinoma (RCC). A control group was formed by measuring plasma GAGs in healthy volunteers. The primary endpoints were the specificity and sensitivity of plasma GAGs in the detection of early stage RCC in pre-surgical samples versus healthy individuals. The investigators further analyzed how plasma GAGs varied according to stage, grade, RCC histology, other renal masses, and after surgery. Finally, the investigators estimated whether plasma GAGs could be used for prediction and surveillance of RCC recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiographic finding of renal mass referred to primary surgery;
* Healthy volunteers without any history of malignancy.

Exclusion Criteria:

* No records on date of surgery;
* A pre-operative sample was obtained 50 days or earlier with respect to the date of surgery; - Absence of pre-operative samples following filtering out outliers or laboratory assay failures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with pathologically confirmed diagnosis of RCC treated with surgical resection of the tumor
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2016-04-28 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Specificity and sensitivity of plasma GAGs in the detection of low stage RCC in pre-surgical samples versus healthy individuals | 1 month

SECONDARY OUTCOMES:
Pearson correlation coefficient with plasma GAG score in pre-surgical samples and tumor size in cm | 1 month
Shift in plasma GAG score in pre-surgical samples between locally-advanced or advanced vs. localized RCC | 1 month
  The shift is the absolute difference plasma GAG score, which is measured in arbitrary units in the range 0 to +Inf with higher values associated with RCC versus healthy status.
Shift in plasma GAG score in pre-surgical samples between Fuhrman Nuclear Grade 3+ vs. 2 in clear cell RCC. | 1 month
  The shift is the absolute difference plasma GAG score, which is measured in arbitrary units in the range 0 to +Inf with higher values associated with RCC versus healthy status.
Shift in plasma GAG score in pre-surgical samples between clear cell vs. non-clear cell RCC | 1 month
  The shift is the absolute difference plasma GAG score, which is measured in arbitrary units in the range 0 to +Inf with higher values associated with RCC versus healthy status.
Hazard ratio of plasma GAG score dichotomized in "Low" vs. "High" score in pre-surgical samples for overall survival in RCC | 53 months
  The dichotomized plasma GAG score is a categorical binary variable based on a post-hoc cut-off value for the plasma GAG score, which is measured in arbitrary units in the range 0 to +Inf with higher values associated with RCC versus healthy status.
Hazard ratio of plasma GAG score dichotomized in "Low" vs. "High" score in pre-surgical samples for metastatic recurrence-free survival in RCC | 53 months
  The dichotomized plasma GAG score is a categorical binary variable based on a post-hoc cut-off value for the plasma GAG score, which is measured in arbitrary units in the range 0 to +Inf with higher values associated with RCC versus healthy status.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gatto F, Blum KA, Hosseini SS, Ghanaat M, Kashan M, Maccari F, Galeotti F, Hsieh JJ, Volpi N, Hakimi AA, Nielsen J. Plasma Glycosaminoglycans as Diagnostic and Prognostic Biomarkers in Surgically Treated Renal Cell Carcinoma. Eur Urol Oncol. 2018 Oct;1(5):364-377. doi: 10.1016/j.euo.2018.04.015. Epub 2018 Jun 13. PMID 31158075